CLINICAL TRIAL: NCT00160563
Title: The Prolongation of the EPAAC™ Trial - NCT00152464 (The Early Prevention of Asthma in Atopic Children). A Multi-country, Double Blind, Placebo (PLC) Controlled, Follow-up Trial With 3 Parallel Groups (LCTZ-LCTZ, LCTZ-PLC and PLC-PLC) : Evaluation of the Long Term Efficacy and Safety of Levocetirizine (LCTZ) (5 mg/ml Oral Drops -0.125 mg/kg b.w. b.i.d.) Administered for an Additional 18 Months Period in Preventing the Onset of Asthma in Children Coming From the EPAAC Trial.
Brief Title: Prevention of Asthma With Levocetirizine (36 Month Treatment) in Young Children Suffering From Eczema (Atopic Dermatitis) and Sensitized to Grass Pollen and House Dust Mite and Having Completed the Previous EPAAC Trial (NCT00152464)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The predecessor study A00309 (NCT00152464) did not show statistical significance in time to onset of asthma between the levocetirizine and placebo groups.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A00384
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
Keywords: Pediatry; EPAAC; atopic Children; prevention of asthma; Levocetirizine; Xyzal
MeSH Terms: conditions — Asthma | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LCTZ-LCTZ (Experimental): Levocetirizine after having been randomized to Levocetirizine in the preceding A00309 trial - NCT00152464 (LCTZ-LCTZ)
  Interventions: Drug: LEVOCETIRIZINE
- LCTZ-PLC (Placebo Comparator): Placebo after having been randomized to Levocetirizine in the preceding A00309 trial - NCT00152464 (LCTZ - PLC)
  Interventions: Other: Placebo
- PLC-PLC (Placebo Comparator): Placebo after having been randomized to Placebo in the preceding A00309 trial - NCT00152464 (PLC-PLC)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LEVOCETIRIZINE — 5mg/mL oral drops, 0.125 mg/kg body weight, bid for 18 months
  Other Names: Xyzal®
  Arms: LCTZ-LCTZ
Other: Placebo — Oral drops, bid for 18 months
  Arms: LCTZ-PLC; PLC-PLC

SUMMARY:
Prolongation of the EPAAC™ trial - NCT00152464 (The Early Prevention of Asthma in Atopic Children).

36 months study to evaluate the efficacy and safety of levocetirizine (LCTZ) in preventing the onset of asthma in young atopic children.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria which must be verified at the end of first 18-months treatment (Visit 9)

* Having completed the previous 18-month treatment period of the EPAAC trial - NCT00152464

Exclusion Criteria:

* None

Ages: 30 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Campine, MD, Study Director — UCB Pharma
Locations (51):
- Australia (2):
  - North Adelaide
  - Parkville (North Melbourne)
- Brussels, Belgium
- Czechia (6):
  - Brno
  - Hradec Králové
  - Olomouc
  - Ostrava
  - Plezen-Lochotin
  - Prague
- France (4):
  - Martigues
  - Saint-Etienne
  - Tarbes
  - Toulouse
- Germany (8):
  - Bayreuth
  - Berlin
  - Bielefeld
  - Bochum
  - Cologne
  - Erlangen
  - München
  - Wesel
- Italy (8):
  - Ancona
  - Bari
  - Bologna
  - Messina
  - Milan
  - Napoli
  - Pavia
  - Roma
- Poland (8):
  - Bialystock
  - Gdansk
  - Karpacz
  - Lodz
  - Lublin
  - Rabka-Zdrój
  - Warsaw
  - Wroclaw
- South Africa (9):
  - Bellville
  - Clarement
  - Durban
  - Mowbray
  - Pietermaritzburg
  - Sydenham
  - West Honeydew
  - Westville
  - Wynberg
- Spain (2):
  - Barcelona
  - Espluques de Llobreqat
- United Kingdom (3):
  - Dorchester
  - Enfield
  - Southampton

REFERENCES:
- See also: For FDA Safety Alerts and Recalls refer to — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a 18-month prolongation study to study A00309 (EPAAC study - NCT00152464) and was prematurely terminated due to the fact that the primary endpoint in study A00309 - NCT00152464 was not met.
Pre-assignment Details: In total, 207 subjects from study A00309 - NCT00152464 entered this prolongation study. Participants Flow and Baseline Characteristics sections show patients as randomized. One patient (016/1709) received LCTZ instead of PLC in the PLC-PLC arm erroneously and is described separately in the Adverse Event section.
Groups:
- LCTZ-LCTZ: Levocetirizine after having been randomized to Levocetirizine in the preceding A00309 trial (LCTZ-LCTZ)
- LCTZ-PLC: Placebo after having been randomized to Levocetirizine in the preceding A00309 trial (LCTZ - PLC)
- PLC-PLC: Placebo after having been randomized to Placebo in the preceding A00309 trial (PLC-PLC)
Period: Overall Study
Arm/Group | LCTZ-LCTZ | LCTZ-PLC | PLC-PLC
Started | 59 | 47 | 101
Completed | 8 | 2 | 11
Not Completed | 51 | 45 | 90
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 3
Not completed — Other (listed in the study report) | 48 | 40 | 81
Not completed — Missing reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCTZ-LCTZ | LCTZ-PLC | PLC-PLC | Total
Number analyzed (Participants) | 59 | 47 | 101 | 207
Age, Continuous [Mean (Standard Deviation); unit: months] | 19.6 (3.58) | 18.9 (4.08) | 19.2 (4.10) | 19.2 (3.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 38 | 86
  Male | 36 | 22 | 63 | 121
Region of Enrollment [Number; unit: participants]
  France | 2 | 3 | 9 | 14
  Czech Republic | 9 | 8 | 17 | 34
  Poland | 11 | 9 | 18 | 38
  Spain | 0 | 1 | 2 | 3
  Belgium | 3 | 0 | 1 | 4
  Australia | 2 | 3 | 2 | 7
  South Africa | 15 | 10 | 22 | 47
  Germany | 9 | 4 | 13 | 26
  Italy | 6 | 7 | 13 | 26
  United Kingdom | 2 | 2 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Asthma
Time Frame: 36 months (from the randomization visit to the preceding A00309 - NCT00152464 trial onwards.)
Population: Analysis was not performed due to premature discontinuation of the study.
Arm/Group | LCTZ-LCTZ | LCTZ-PLC | PLC-PLC
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Time to Onset of Asthma in the Subset of Subjects Still Asthma Free After First 18 Months.
Time Frame: 18 months (from the end of the preceding A00309 - NCT00152464 trial onwards.)
Population: Analysis was not performed due to premature discontinuation of the study.
Arm/Group | LCTZ-LCTZ | LCTZ-PLC | PLC-PLC
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- PLC-LCTZ: Levocetirizine after having been randomized to Placebo in the preceding A00309 trial (PLC-LCTZ) erroneously (Patient 016/1709)
Arm/Group | LCTZ-LCTZ | LCTZ-PLC | PLC-PLC | PLC-LCTZ
Serious Adverse Events (participants affected / at risk) | 5/59 | 3/47 | 3/100 | 0/1
Other Adverse Events (participants affected / at risk) | 48/59 | 36/47 | 71/100 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCTZ-LCTZ (N=59) | LCTZ-PLC (N=47) | PLC-PLC (N=100) | PLC-LCTZ (N=1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCTZ-LCTZ (N=59) | LCTZ-PLC (N=47) | PLC-PLC (N=100) | PLC-LCTZ (N=1)
Conjunctivitis (Eye disorders) | 3 (4) | 5 (8) | 5 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 4 (6) | 5 (6) | 0 (0)
Pyrexia (General disorders) | 10 (13) | 7 (9) | 13 (20) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 4 (5) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 9 (11) | 6 (10) | 16 (26) | 0 (0)
Bronchitis acute (Infections and infestations) | 3 (5) | 3 (4) | 5 (6) | 0 (0)
Ear infection (Infections and infestations) | 5 (7) | 2 (3) | 6 (10) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (10) | 2 (2) | 9 (11) | 0 (0)
Laryngitis (Infections and infestations) | 4 (5) | 3 (4) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (15) | 11 (21) | 17 (46) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 4 (5) | 9 (15) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (2) | 5 (6) | 0 (0)
Pharyngitis (Infections and infestations) | 8 (10) | 10 (27) | 12 (19) | 0 (0)
Rhinitis (Infections and infestations) | 15 (32) | 3 (4) | 12 (32) | 1 (1)
Scarlet fever (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (3) | 1 (2) | 10 (11) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (46) | 10 (30) | 20 (48) | 0 (0)
Varicella (Infections and infestations) | 3 (3) | 2 (2) | 7 (7) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 5 (6) | 4 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.